CLINICAL TRIAL: NCT01706770
Title: Evaluation of Enfilcon A Soft Contact Lens Compared to Galyfilcon A Soft Contact Lens
Brief Title: Evaluation of Enfilcon A Soft Contact Lens When Compared to Galyfilcon A Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FC111216
Record Dates: First submitted 2012-10-05; First posted 2012-10-15 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- enfilcon A (Experimental): The test (experimental) lens is a silicone hydrogel contact lens following a daily wear 1 week planned replacement modality.
  Interventions: Device: enfilcon A
- galyfilcon A (Active Comparator): The control (active comparator) lens is a silicone hydrogel contact lens following a daily wear 1 week planned replacement modality.
  Interventions: Device: galyfilcon A

INTERVENTIONS:
Device: enfilcon A
  Other Names: Avaira® Toric
  Arms: enfilcon A
Device: galyfilcon A
  Other Names: Acvuve® Advance®
  Arms: galyfilcon A

SUMMARY:
The primary objective of thes study is to confirm that the ocular response to the Test lenses are similar to those of the Control lenses when used in a 1 week planned replacement, daily wear modality over a 1-month period.

DETAILED DESCRIPTION:
The test lens and control lens were randomized in a 2:1 ratio to evaluate the test lens and control contact lens.

ELIGIBILITY:
Inclusion Criteria:

Prior to being considered eligible to participate in this study, each subject MUST:

* Be at least 18 years of age as of the date of evaluation for the study.
* Have read the Informed Consent, been given an explanation of the Informed Consent, indicated understanding of the Informed Consent, signed the Informed Consent document.
* Be willing and able to adhere to the instructions set forth in this protocol and able to keep all specified appointments.
* Be an adapted, current full-time silicone hydrogel or soft contact lens wearer. An adapted full-time wearer is defined as wearing contact lenses in both eyes on a daily basis for at least 8 hours per day for at least one month prior to participation in the study.
* Possess wearable and visually functional eyeglasses.
* Be in good general health, based on his/her knowledge.
* Require spectacle lens powers between -1.00 and -6.00 diopters sphere with no more than 2.00 diopters of refractive astigmatism and be willing to wear contact lenses in both eyes.
* Have: manifest refraction Snellen visual acuities (VA) equal to or better than 20/25 in each eye.
* Upon completing the fitting process with the lenses to be worn in the study, have contact lens Snellen VA equal to or better than 20/30 in each eye.

Exclusion Criteria:

Subjects may not be enrolled in this study if any of the following apply: The subject is/has:

* Wearing lenses in a monovision modality and is unwilling to be fit with distance lenses in both eyes. NOTE: Subjects may not wear lenses in a monovision modality at any time during the study as it will interfere with the visual acuity analysis.
* Poor personal hygiene.
* Any active participation in another clinical trial within 30 days prior to this study.
* Currently pregnant (to the best of the subject's knowledge), is lactating or is planning a pregnancy within the study period.
* A member, relative or household member of the investigator or of the investigational office staff.
* Has a known sensitivity to ingredients used in the care products approved for use in the study.
* Previous refractive surgery; or current or previous orthokeratology treatment.
* Is aphakic or psuedophakic.
* Ocular or systemic disease such as, but not limited to: anterior uveitis or iritis (past or present), glaucoma, Sjögren's syndrome, lupus erythematosus, sclerodermia, keratoconus or type II diabetes.
* The need for topical ocular medications or any medication which might interfere with contact lens wear or which would require the lenses to be removed during the day.
* The presence of clinically significant (grade 3 or 4) anterior segment abnormalities.
* Any; inflammations such as iritis; or any infection or allergic reaction of the eye, lids, or associated structures.
* A known history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates or fungal infections.
* A history of papillary conjunctivitis that has interfered with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear, including but not limited to: Pathological dry eye or associated dry eye symptoms with decreased tear levels and punctuate staining > Grade 2, Pterygium, Corneal scars within the visual axis, Neovascularization or ghost vessels > 1.0 mm in from the limbus, Giant papillary conjunctivitis (GPC) of > Grade 1, Anterior uveitis or iritis, Seborrheic eczema, seborrheic conjunctivitis or blepharitis

To be eligible to be randomized for study product a subject must have ALL of the Inclusion Criteria and have NONE of the exclusion criteria present.

To be eligible for lens dispensing (either Test or Control), the subject's study lens contact lens visual acuity must be equal to or better than 20/30 in each eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Schachter, OD, Principal Investigator — Unafiliated; Cheryl Vincent-Reimer, OD, Principal Investigator — Unafiliated; Eric White, OD, Principal Investigator — Unafiliated
Locations (3):
- United States (3):
  - Advanced Eyecare, Pismo Beach, California
  - Eric M. White, OD, Inc., San Diego, California
  - Vision Care Associates, East Lansing, Michigan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 52 subjects evaluated. Of these 52 subjects, 2 found ineligible and not randomized resulting in 50 subjects randomized, 33 test, 17 control. Of 50 subjects randomized, 2 discontinued and not included in results data, 31 test, 17 control, 1 lost to follow-up, 1 Sponsor/IRB decision due to pregnancy at one month visit.
Period: Overall Study
Arm/Group | Enfilcon A | Galyfilcon A
Started | 33 | 17
Completed | 31 | 17
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enfilcon A | Galyfilcon A | Total
Number analyzed (Participants) | 33 | 17 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 17 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (11.11) | 33.8 (11.50) | 34.4 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 12 | 35
  Male | 10 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 33 | 17 | 50

OUTCOME MEASURES:

1. Primary Outcome: Objective Assessment: Ocular Response - Biomicroscopy
Description: The primary safety endpoint are the objective slit lamp findings associated with the enfilcon A contact lenses compared with those same findings reported as associated with the galyfilcon A contact lenses.
  The incidence of biomicroscopy findings (0=not present, 4=severe) over the duration of the study with the highest reported grade was chosen for each unique eye. Biomicroscopy measurements were obtained at Baseline/Dispensing (baseline and dispensing visit combined), Post-Dispensing (after lenses were dispensed and allowed to settle) and All Follow-Ups (week 1 visit, week 2 visit, month 1 visit combined). The average grade for unique eyes with findings greater than 0 (none) is compared.
Time Frame: Change from baseline/dispensing visits, post-dispensing visit and all follow-ups visits
Population: Unique eyes are defined as each individual eye in the study and are only counted once for each of the visit groupings.
Measure: Mean (Full Range); unit: units on a scale
Units Other Than Participants: unique eyes
Arm/Group | Enfilcon A | Galyfilcon A
Number analyzed (Participants) | 31 | 17
Number analyzed (unique eyes) | 62 | 34
units on a scale
  Epithelial Edema, Baseline/Dispensing | 1.00 [1 to 1] | NA [0 to 0] — No participants experienced greater than 0 at this time point.
  Epithelial Edema, Post-Dispensing | NA [0 to 0] — No participants experienced greater than 0 at this time point. | NA [0 to 0] — No participants experienced greater than 0 at this time point.
  Epithelial Edema, All Follow-up | NA [0 to 0] — No participants experienced greater than 0 at this time point. | NA [0 to 0] — No participants experienced greater than 0 at this time point.
  Stromal Edema, Basline/Dispensing | NA [0 to 0] — No participants experienced greater than 0 at this time point. | NA [0 to 0] — No participants experienced greater than 0 at this time point.
  Stromal Edema, Post-Dispensing | NA [0 to 0] — No participants experienced greater than 0 at this time point. | NA [0 to 0] — No participants experienced greater than 0 at this time point.
  Stromal Edema, All Follow-up | NA [0 to 0] — No participants experienced greater than 0 at this time point. | NA [0 to 0] — No participants experienced greater than 0 at this time point.
  Neovascularization, Baseline/Dispensing | 1.00 [1 to 1] | 1.00 [1 to 1]
  Neovascularization, Post-Dispensing | NA [0 to 0] — No participants experienced greater than 0 at this time point. | 1.00 [1 to 1]
  Neovascularization, All Follow-up | 1.00 [1 to 1] | 1.00 [1 to 1]
  Corneal Staining, Baseline/Dispensing | 1.06 [1 to 2] | 1.08 [1 to 2]
  Corneal Staining, Post-Dispensing | 1.00 [1 to 1] | 1.00 [1 to 1]
  Corneal Staining, All Follow-up | 1.02 [1 to 2] | 1.04 [1 to 2]
  Limbal Hyperemia, Baseline/Dispensing | 1.07 [1 to 2] | 1.00 [1 to 1]
  Limbal Hyperemia, Post-Dispensing | 1.00 [1 to 1] | 1.00 [1 to 1]
  Limbal Hyperemia, All Follow-up | 1.00 [1 to 1] | 1.00 [1 to 1]
  Bulbar Hyperemia, Baseline/Dispensing | 1.00 [1 to 1] | 1.00 [1 to 1]
  Bulbar Hyperemia, Post-Dispensing | 1.00 [1 to 1] | 1.00 [1 to 1]
  Bulbar Hyperemia, All Follow-up | 1.00 [1 to 1] | 1.00 [1 to 1]
  Palpebral Conjunctiva, Baseline/Dispensing | 1.11 [1 to 2] | 1.12 [1 to 2]
  Palpebral Conjunctiva, Post-Dispensing | 1.00 [1 to 1] | 1.14 [1 to 2]
  Palpebral Conjunctiva, All Follow-up | 1.05 [1 to 2] | 1.16 [1 to 2]

2. Primary Outcome: Comparison of Objective Findings - Number of Adverse Events in Unique Eyes
Description: The primary safety endpoint are the objective findings of the number of adverse events in unique eyes associated with the enfilcon A contact lenses compared with those same findings as associated with the galyfilcon A contact lenses.
  The number of adverse events over the duration of the study was reported for each unique eye (bilateral or unilateral). Observations for adverse events were reported for any occurrence from Baseline through end of month 1 visit.
Time Frame: Any occurrence from baseline to 1 month visit
Population: Unique eyes are defined as each individual eye in the study.
Measure: Number; unit: number of adverse events
Units Other Than Participants: eyes
Arm/Group | Enfilcon A | Galyfilcon A
Number analyzed (Participants) | 31 | 17
Number analyzed (eyes) | 62 | 34
number of adverse events | 0 | 2

ADVERSE EVENTS:
Time Frame: From dispense up to one month on both the study lenses, a total of two months.
Arm/Group | Enfilcon A | Galyfilcon A
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/17
Other Adverse Events (participants affected / at risk) | 0/33 | 1/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enfilcon A (N=33) | Galyfilcon A (N=17)
Temporary Discontinuation of Lens Wear (Eye disorders) | 0 (0) | 1 (1) — Single (one subject), bilateral event reported for the control group at day 21 as temporary discontinuation lens wear of 1 day. Subject napped with lenses in place. Awoke with red eyes. Removed the lenses for the remainder of the day.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Release of this data (through presentation, publication or other written or oral communication) to other than listed personnel (see protocol) requires the prior written permission from the study Sponsor. Study investigators and all office personnelare prohibited from acknowledging participation in the study to individuals and organizations except those listed.